CLINICAL TRIAL: NCT04251312
Title: Minimizing Pathologic Aspiration in Patients Undergoing Esophageal and Lung Resections for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Jacob Moremen, Assistant Professor of Cardio-Thoracic Surgery, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0327
Record Dates: First submitted 2020-01-16; First posted 2020-01-31 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Cancer; Lung Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative dental hygiene education (Experimental): Patients who are scheduled for elective esophageal or lung resections who consent to participate will undergo oral hygiene education and be given an oral hygiene packet. An oral hygiene assessment using the Plaque Assessment tool will be conducted in the clinic. A Dysphagia Screening Tool questionnaire will also be administered. Patients who screen positive for dysphagia will be referred to Speech Pathology for evaluation but for the study purposes, the only data collected from the evaluation will be whether or not the participant received this intervention. A repeat dental exam will occur on the day of surgery. Patients will be followed for 30 days post operatively.
  Interventions: Other: Oral Hygiene Education and Oral Hygiene Packets

INTERVENTIONS:
Other: Oral Hygiene Education and Oral Hygiene Packets — Patients will be educated on oral hygiene and will be given packets containing toothpaste, mouth rinse, floss and a toothbrush

SUMMARY:
The aim of this study is to reduce pathologic aspiration and pneumonia in the perioperative period by providing an oral care and oral hygiene education to patients preoperatively. Patients enrolled in the study will be given a dysphagia screening questionnaire, an oral care package and oral hygiene education. Patients who screen positive for dysphagia will be referred to Speech Pathology for evaluation. The rate of postoperative pneumonia will be determined for those who participate in the study and will be compared to retrospective patient data from our institution.

DETAILED DESCRIPTION:
Aspiration by high risk esophageal and lung cancer patients with either preexisting or post-therapy/post-operative dysphagia leads to morbidity (pneumonia) and mortality following surgery. The aim of this study is to reduce pathologic aspiration and pneumonia in the perioperative period by providing an oral care and oral hygiene education to patients preoperatively. Patients enrolled in the study will be given a dysphagia screening questionnaire, an oral care package and oral hygiene education. Patients who screen positive for dysphagia will be referred to Speech Pathology for evaluation. The rate of postoperative pneumonia will be determined for those who participate in the study and will be compared to retrospective patient data from our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective esophageal or lung resections for cancer at our institution

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Proportion of pneumonia | 6 months
  Number of participants who develop postoperative pneumonia in the interventional arm compared to the number of patients retrospectively reviewed who received no intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Moremen, M.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
After appropriate consent, patient charts will be reviewed by study members that have completed appropriate training. Protected Health Information (PHI) that will be accessed includes demographic data for patients such as Medical Record Number, date of surgery, planned operation, dental history, etc.(Also see the Data Collection Form). PHI will be collected and maintained in REDCap. For the retrospective review portion of the study, the charts of previous patients will be accessed. Data from those patients who underwent surgery within one year prior to beginning the study will be compared to the data collected during the study. Since obtaining consent for this portion of chart review will be difficult, we plan to request a HIPAA waiver of authorization.

REFERENCES:
- [Result] Semenkovich TR, Frederiksen C, Hudson JL, Subramanian M, Kollef MH, Patterson GA, Kreisel D, Meyers BF, Kozower BD, Puri V. Postoperative Pneumonia Prevention in Pulmonary Resections: A Feasibility Pilot Study. Ann Thorac Surg. 2019 Jan;107(1):262-270. doi: 10.1016/j.athoracsur.2018.08.008. Epub 2018 Oct 3. PMID 30291834
- [Result] Soutome S, Yanamoto S, Funahara M, Hasegawa T, Komori T, Yamada SI, Kurita H, Yamauchi C, Shibuya Y, Kojima Y, Nakahara H, Oho T, Umeda M. Effect of perioperative oral care on prevention of postoperative pneumonia associated with esophageal cancer surgery: A multicenter case-control study with propensity score matching analysis. Medicine (Baltimore). 2017 Aug;96(33):e7436. doi: 10.1097/MD.0000000000007436. PMID 28816937
- [Result] Hernan MA, Robins JM. Estimating causal effects from epidemiological data. J Epidemiol Community Health. 2006 Jul;60(7):578-86. doi: 10.1136/jech.2004.029496. PMID 16790829